CLINICAL TRIAL: NCT07278648
Title: Prescription of High-risk Antithrombotic Drugs at Discharge and Consultation for Hemorrhagic or Thromboembolic Events in the Emergency Department. Retrospective Cohort Study
Brief Title: High-risk Antithrombotic Drugs at Discharge and Consultation for Hemorrhagic or Thromboembolic Events in the Emergency Department
Status: Not yet recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-79
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Disease
Keywords: Antithrombotic Treatment; Hemorragic Event; Anticoagulants
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anticoagulant therapy: Patients who has been discharged from hospital with anticoagulant therapy
  Interventions: Other: Antithrombotic therapy

INTERVENTIONS:
Other: Antithrombotic therapy — Anticoagulant treatment prescribed at discharge from an acute care unit

SUMMARY:
This observational study aims to estimate the proportion of patients discharged from a hospital with a prescription for anticoagulant medication who subsequently visit the emergency department due to an adverse thrombotic or hemorrhagic event related to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from the Emergency Department (ED) and acute care units with an electronic prescription for at least one anticoagulant medication (new or ongoing), identified with the following codes:

B01AA - Vitamin K antagonists: warfarin and acenocoumarol

B01AB - Heparin group: low-molecular weight heparins such as enoxaparin, tinzaparin, bemiparin, …

B01AE - Direct thrombin inhibitors: dabigatran

B01AF - Direct factor Xa inhibitors: rivaroxaban, apixaban, edoxaban

Exclusion Criteria:

* Those who are not part of the CSAPG healthcare area.
* Patients discharged from outpatient clinics, home hospitalization units, intermediate care, or residential facilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who has been discharged from an acute care unit with anticoagulant therapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Hemorragic event | Day 90 from baseline
  Proportion of patients who experience a hemorrhagic event within 90 days of hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Vilafranca, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.